CLINICAL TRIAL: NCT02942784
Title: Prediction of Prognosis in Patients With Chronic Obstructive Pulmonary Disease With Respiratory Failure: A Comparison of Three Nutritional Assessment Methods
Brief Title: A Comparison of Three Nutritional Assessment Methods Predicting Prognosis in COPD With Respiratory Failure
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lu Xing, Principal Investigator, Master Degree, West China Hospital
Other Study IDs: COPD-001
Record Dates: First submitted 2016-10-10; First posted 2016-10-24 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective study of patients diagnosed with chronic obstructive pulmonary disease (COPD) with respiratory failure and admitted in West China Hospital during January 2014 to March 2016 by review of medical records. The following variables will be retrospectively studied: age, sex, marriage, height, weight, respiratory rate, PaO2, PaCO2, nutritional risk screening 2002 (NRS 2002) score, ALB, short-term and long-term prognostic outcomes, and so on. The purpose of this study is to compare the predictive power of three widely used nutritional assessment methods (BMI, NRS 2002 and ALB) predicting the prognostic outcomes in a cohort of COPD patients with respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis of COPD at West China Hospital during January 2014 to March 2016
* Partial pressure of O2 (PaO2) < 60 mmHg and/or partial pressure of CO2 (PaCO2) >50 mmHg
* Age ≥ 18 years
* Respiratory rates > 23 bpm

Exclusion Criteria:

* Pregnancy or during lactation
* Ventilatory dysfunction due to neuromuscular disorders, acute and chronic thromboembolic disease, severe illness in other systems
* Incomplete medical profiles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with chronic obstructive pulmonary disease with respiratory failure during January 2014 to March 2016 at West China Hospital by review of medical records.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Predictive value of nutritional assessment methods in identifying COPD patients with respiratory failure who will have poor prognosis, in terms of in-hospital death | up to 27 months
Predictive value of nutritional assessment methods in identifying COPD patients with respiratory failure who will have poor prognosis, in terms of 1-year death after discharge | up to 27 months
Predictive value of nutritional assessment methods in identifying COPD patients with respiratory failure who will have poor prognosis, in terms of 30-day readmission after discharge | up to 27 months

SECONDARY OUTCOMES:
Collection of Demographics (age, sex, marriage) | up to 27 months
Number of participants with in-hospital death | up to 27 months
Number of participants with 1-year death after discharge | up to 27 months
Number of participants with 30-day readmission after discharge | up to 27 months

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China